CLINICAL TRIAL: NCT02916628
Title: Effects of Auricular Acupressure and Group Therapy on Smoking Cessation Tobacco Withdrawal Symptoms, Depressive Symptoms, Resilience, and Serum Serotonin Level
Brief Title: Effects of Auricular Acupressure and Group Counseling on Smoking Cessation Tobacco Withdrawal Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, EUN JIN LEE, Associate professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-03-058
Record Dates: First submitted 2016-09-20; First posted 2016-09-27 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Smoking
Keywords: smoking cessation; group counseling; acupressure; serotonin; depressive symptoms; resilience
MeSH Terms: conditions — Smoking; Smoking Cessation; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): auricular acupressure + group counseling
  Interventions: Behavioral: group counseling; Device: Auricular acupressure
- Group 2 (Placebo Comparator): placebo acupressure + group counseling
  Interventions: Behavioral: group counseling; Device: placebo acupressure
- Group 3 (No Intervention): self-help smoking cessation
- Group 4 (No Intervention): Non-smokers

INTERVENTIONS:
Behavioral: group counseling — Group counseling with positive psychology and motivational interviewing was undertaken once per week for 6 weeks.
  Arms: Group 1; Group 2
Device: Auricular acupressure — Auricular acupressure using acupellets was performed for 6 weeks continuously
  Arms: Group 1
Device: placebo acupressure — Placebo acupellets were prepared without metal projections, and placed on both sides in the same areas of the ear as the active condition.
  Arms: Group 2

SUMMARY:
Objective The purpose of this study is to examine the effects of auricular acupressure and group counseling with positive psychology and motivational interviewing on smoking cessation and tobacco withdrawal symptoms.

Methods This study is a single blind randomized controlled trial. This study has been performed at a University in South Korea. 180 smokers and 60 non-smokers will be recruited. Smokers will be randomly assigned to three groups: group 1 (auricular acupressure + group counseling); group 2 (placebo acupressure + group counseling); and the control group (self-help smoking cessation). Group counseling is undertaken once per week for 6 weeks. Auricular acupressure using acupellets is performed for 6 weeks continuously.

DETAILED DESCRIPTION:
1. Introduction South Korea takes second place for its smoking rate among 22 member countries in the Organization for Economic Co-operation and Development (OECD). The smoking rate in the U.S. is 16.8% among adults aged 18 years or older, while the smoking rate in South Korea is 42.6%. Medical costs spent on diseases caused by smoking are estimated to be 1.53 billion dollars, accounting for 3.7% of all health insurance medical costs spent in 2012 in South Korea. In 2010, 54.9% of smokers tried to quit smoking. Concerns about health accounted for 67.7% of the motivation for smoking cessation. Compared to non-smoking men, male smokers have a 6.5, 4.6, and 3.6 fold increased risk of getting cancer of the larynx, lungs, and esophagus, respectively. Of smokers who tried to quit smoking, 84.7% did not have any assistance. Smokers reported that main reasons for failing smoking cessation were stress and withdrawal symptoms.

   To increase the success rate in smoking cessation, stress management and reduction of withdrawal symptoms are very important. Many methods have been used to assist smoking cessation. These methods include cognitive behavioral therapy, antidepressants, nicotine patches, nicotine gum, positive psychology, motivational interviewing, acupuncture, and acupressure. Traditional psychiatric approaches focus on what is wrong, while positive psychology focuses on strength and values that empower individuals. Positive psychology deals with stress management using gratitude, love, forgiveness, and hope. Motivational interviewing is a "directive client-centered counseling approach for initiating behavior change by helping clients to resolve ambivalence". Acupuncture uses needles to stimulate acupuncture points, while acupressure uses fingers, hands, beads, or pellets to stimulate acupuncture points. Stimulation of acupuncture points reduces withdrawal symptoms by reducing desire or changing tastes. The mechanism of acupuncture on smoking cessation has not examined well. Cabioglu and his colleagues suggested that acupuncture may increase the levels of several neurotransmitters such as dopamine and serotonin.

   There is no consistent evidence that acupuncture is effective for smoking cessation. Tahiri and his colleagues reported the smoking rate of acupuncture was 3%-55% at 6-month follow-ups based on 6 randomized controlled trials. Authors have suggested more randomized controlled studies are needed. A few studies have examined the effect of positive group psychotherapy on smoking cessation. In addition, only a few studies have examined the mechanism of acupressure on smoking cessation.

   The purpose of this study was to examine the effects of auricular acupressure and group counseling with positive psychology and motivational interviewing on smoking cessation and reduction, tobacco withdrawal symptoms, depressive symptoms, and serum serotonin levels.
2. Methods 2.1. Design and setting The design of this study is a single blind randomized controlled trial. This study will be conducted at a University in South Korea from July 2013 to July 2017.

2.2. Sample selection Smokers will be recruited by internet advertisement or face-to-face contacts. All smokers were informed about the study protocol, benefits and side effects of interventions, and the right to withdraw from the study at any time without penalty. Smokers who agree to participate in this study signed consent forms before data collection. Ethical approval was obtained from the institutional review board in Incheon, South Korea.

2.3. Randomization and single blinding Randomization of numbers was done by random.org. Opaque envelopes with numbers are prepared and participants drew numbers from a container. Participants will be randomly assigned to one of three groups: group 1 (auricular acupressure + group counseling); group 2 (placebo acupressure + group counseling); or the control group (self-help smoking cessation). The researcher will give participants envelopes with questionnaires to complete. Participants put the questionnaires into the envelope after completion. Groups 1 and 2 do not know about their allocation. The researcher does not know about the results of the questionnaires before the completion of the study. The research assistants will perform coding on the questionnaire data.

2.4. Procedure All participants set a quit date for one week from enrollment in the study. Information for reducing withdrawal symptoms will be provided to all participants. Groups 1 and 2 will be instructed not to stimulate themselves with acupellets. They will be informed that acupellets would be changed every week, even if the acupellets fell off before the next appointment. Group counseling and acupressure will be performed by the researcher, who is a psychiatric-mental health nurse practitioner and an acupuncturist. Group counseling consisted of positive psychology and motivational interviewing. Each group consisted of 3-5 participants. Group 1 will receive group counseling for one hour per week for 6 weeks. At the beginning of each group psychotherapy session, participants talked about the number of cigarettes smoked during the previous week, and any coping methods used to maintain abstinence or to reduce smoking.

Auricular acupressure with acupellets will be performed by the researcher at a relaxation point, lung point, nicotine point, thirst point, and antidepressant point on both sides, once per week for 6 weeks. Acupellets are stickers that have copper or aluminum projections. If participants will report an allergy to copper, then acupellets with aluminum projections will be applied; if participants reported an allergy to aluminum, then acupellets with copper projections were applied. If prospective participants are allergic to both copper and aluminum, then they will be excluded from the study. Group 2 will receive positive group psychotherapy 1 hour per week for 6 weeks. Placebo acupellets will be prepared without metal projections, and placed on both sides in the same areas of the ear as the active condition. Auricular acupressure using acupellets will be performed for 6 weeks continuously. Group counseling and auricular acupressure will be undertaken at the same time. The control group will be encouraged to quit smoking without acupressure and psychotherapy. If the control group cannot quit smoking after 6 weeks, participants in the control group will then instructed to apply acupellets at the same five auricular acupressure sites as previously described. A picture of ears with acupressure points will be provided.

2.5. Data collection At baseline, all participants completed demographic and smoking-related questions, and the Patient Health Questionnaire (PHQ)-9. Participants will complete the Minnesota Tobacco Withdrawal Scale (MTWS) during the 6-week period. Urine cotinine tests will perform at 6 weeks, 6 months, and 1 year if participants report that they quit smoking for at least 1 week. Smoking amounts will be assessed five times: at baseline, 6 weeks, 3 months, 6 months, and 1 year. The PHQ-9 and serum serotonin will be assessed at baseline, 6 weeks, 6 months, and 1 year.

2.6. Success of Blinding After 6 weeks, participants in groups 1 and 2 will be asked to which group they think they had been assigned to.

2.7. Sample size calculation and statistical analysis G power was used to calculate sample size. Wu and his colleagues reported the effect size of acupuncture on smoking cessation at the 6-week follow-up was 20.9% ± 7 (n = 64) for group 1 and 17.9% ± 7 (n = 61) for the control group. The effect size using Hedges' g was 0.43 but 0.25 was used because the effect of acupressure was less than acupuncture. Repeated measure ANOVA, within-between interaction, effect size of 0.25, power of 95%, alpha error of 0.05, number of groups 3, number of measurements 4, and correlation among measurements at 0.5 were used. Repeated measure ANOVA will be used because smoking amount, 5-hydroxytryptamine levels, and depression will be measured at four time points and nicotine withdrawal symptoms will be measured at six time points. G power showed that 45 participants will be needed. Statistical Package for the Social Sciences (SPSS) 21.0 will be used for statistical analysis. Normal distribution and homogeneity of variance will be tested. The 5% level of significance and two-tailed test will be used. Intention-to-treat analysis will be used. Missing data were replaced with the previous data. Repeated measures of ANOVA will be used to compare withdrawal symptoms between two groups over 6 weeks. A t-test will be used to compare smoking cessation rates after the intervention between groups. The standard error for the difference of two proportions will be calculated using a formula = square root {[p1 * (1 - p1) / n1] + [p2 * (1 - p2) / n2]}.

ELIGIBILITY:
Inclusion Criteria:

* smokers who:

  1. were more than 19 years
  2. could complete questionnaires
  3. have smoked longer than 6 months
  4. wanted to quit smoking cigarettes
  5. did not have an infection on the surface of the ears.

Exclusion Criteria:

* smokers who

  1. were using nicotine patches or medications for smoking cessation
  2. had allergies to copper or aluminum
  3. had used illegal drugs
  4. were pregnant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
smoking cessation: Change from Baseline Smoking status at 3,6 months, 1 year, 2 years | baseline, 6 weeks, 3 months, 6 months, 1 year, 2 years
  self-report
Minnesota Tobacco Withdrawal Scale(MTWS):Change from Baseline tobacco withdrawal symptoms at 2,3,4,5,6 weeks | baseline,2,3,4,5,6 weeks
  The MTWS was developed to measure nicotine withdrawal symptoms [22]. The MTWS consists of nine items with a 4-point Likert scale. Higher scores indicate more severe withdrawal symptoms. Cronbach's alpha was .88 in 118 Korean Americans. Factor analysis showed two factors: mental difficulties and physical difficulties. These two factors explained 66% of the variance
multidimensional coping scale: Change from Baseline coping skills at 6 weeks, 6 months, 1 year, 2 years | baseline, 6 weeks, 6 months, 1 year, 2 years
  The multidimensional coping scale was developed by Jeon, KG(1994). It consists 50 items including personal, social, and religious coping. The multidimensional coping scale is composed of personal, social, and religious coping resources: (Personal Coping Resources), active coping, passive withdrawal, emotional expression, active forgetting, perseverance, positive interpretation, positive comparison, accommodation, fatalism, self-criticism, emotional pacification; (Social Coping Resources), problem-solving social support seeking, emotional social support seeking; (Religious Coping Resources), religious seeking.
urine cotinine test:Change from 6-week urine cotinine at 6 months, 1 year, 2 years | 6 weeks, 6 months, 1 year, 2 years
  Cotinine is the first-stage metabolite of nicotine. The urine cotinine test using a fresh urine specimen was used to check smoking cessation. There was neither any benefit for smoking cessation in this study nor any legal problem to smoking cigarettes in South Korea. Therefore, participants were allowed to provide urine specimens without close monitoring. The urine cotinine test is a rapid, one-step, immunochromatographic assay for the qualitative detection of cotinine in human urine at 200 ng/ml cut-off concentration. Three drops of urine were transferred to the urine cotinine test apparatus (Brand name: Lungene one step rapid test, Company: Hangzhou Clongene Biotech Co., Ltd, made in China). Two lines indicated a negative result, while one line indicated a positive result. For participants who did not smoke for at least one week, negative test results were expected. Urine cotinine was checked at the 6-week post-test and 6-month follow-up.
serum cotinine levels:Change from 6-week serum cotinine levels at 6 months, 1 year, 2 years | 6 weeks, 6 months, 1 year, 2 years
  Serum cotinine levels reflect recent exposure to nicotine in tobacco smoke. Nonsmoking is usually defined as a serum cotinine level of less than or equal to 10 ng/mL (Pirkle et al., 1996).

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | 6 weeks, 6 months, 1 year, 2 years
  The PHQ-9 was developed to screen for depression. The PHQ-9 consists of nine items with a 4-point Likert scale, which was aligned with diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Higher scores reflect greater depression. Scores suggest no appreciable depression (< 5), mild depression (5-9), moderate depression (10-14), or major depression (≥ 15) [20]. Convergent validity with the Hospital Anxiety Depression Scale was .72 (Pearson correlation coefficient) [21]. Cronbach's alpha was .90 in 193 patients with coronary artery disease.
Resilience | 6 weeks, 6 months, 1 year, 2 years
  The Resilience Scale was developed for children with chronic diseases to measure their capacity to recover quickly from difficulties (D. H. Kim & Yoo, 2010). Lee revised this questionnaire for adolescents (Lee & Cranford, 2008). The Adolescent Resilience Scale consists of 31 items on a 4-point Likert scale. Higher scores reflect strong resilience. Cronbach's α was .93 in 482 adolescents (D. H. Kim & Yoo, 2010). The resilience scale had a significant positive correlation with the Numerical Rating Score and negative correlation with the Child Depression Inventory in 202 children with chronic diseases (r = .51, p<.001; r = -.60, p<.001)
Serum serotonin | 6 weeks, 6 months, 1 year, 2 years
  Five milliliters of blood were drawn from all participants. Blood samples were left at room temperature for 30 minutes for clotting. Blood samples were centrifuged at 3000 rounds per minutes(RPM) for 10 minutes. At least 1 ml of separate serum was collected using a separator. Serum serotonin were kept under -70°C (-94°F). High Performance Liquid Chromatography was used to measure serum serotonin. The Serotonin Kit was made according to Recipe, Germany. Normal range is 101-283 ng/mL
Eysenck Personality Inventory | baseline
  Eysenck Personality Questionnaire (EPQ) is a questionnaire to assess the personality traits of a person, with the result sometimes referred to as the Eysenck's personality Inventory.
  It was devised by the psychologists Hans Jürgen Eysenck and Sybil B. G. Eysenck.
  Hans Eysenck's theory is based primarily on physiology and genetics.

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided